CLINICAL TRIAL: NCT01695122
Title: Efficacy Evaluation of the Combination of Valproic Acid and Standard Platinum-based Chemoradiation in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Valproic Acid and Platinum-based Chemoradiation in Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Milena Mak, MD, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 327/11
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer; Oral Cavity Cancer; Oropharyngeal Cancer
Keywords: Head and Neck Cancer; Oropharyngeal cancer; Oral cavity cancer; Chemoradiation; valproic acid; histone deacetylase
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valproic acid (Experimental)
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid
  Other Names: sodium valproate

SUMMARY:
The purpose of this study is to evaluate if the addition of valproic acid to standard platinum-based chemoradiation as definitive treatment of locally advanced Head and Neck squamous cell carcinoma can improve treatment outcomes, such as response rate.

DETAILED DESCRIPTION:
Valproic acid is a known histone deacetylase inhibitor. In addition to activating apoptosis pathways, cell differentiation and downregulating expression of growth factors, it also promotes radiosensitization.

Most patients with Head and Neck squamous cell carcinoma are diagnosed with locally advanced disease, in which long term disease control is still a challenge. The incorporation of epigenetic regulation into standard treatment could improve results of definitive platinum-based chemoradiation in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable Oropharyngeal or oral cavity squamous cell carcinoma
* Candidate for definitive chemoradiation
* No previous treatment
* Measurable disease according to RECIST v 1.1
* Previous neoplasia, other than Head and Neck, with more than five years without evidence of disease; basocellular carcinoma of the skin and in situ cervical dysplasia if resected
* Age under 60 years
* ECOG performance status 0-2
* Ability of understanding and giving informed consent
* Adequate renal and hepatic function
* Adequate bone marrow function
* Normal serum magnesium
* Absence of QTc prolongation
* Life expectancy of over 12 weeks

Exclusion Criteria:

* Pregnancy
* Distant metastasis
* Hypersensibility to valproic acid or other antiepileptic drugs
* Valproic acid chronic use
* Severe neurologic impairment
* Uncontrolled comorbidity
* Hypoalbuminemia
* Known history of hepatitis B, C or HIV

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Response Rate | Within 6 to 8 weeks after completion of chemoradiation
  RECIST v 1.1

SECONDARY OUTCOMES:
Adverse reactions to study treatment
Progression free survival | Three years
Overall survival | Three Years
Response rate comparison by p16 status
Quality of life

OTHER OUTCOMES:
Biomarkers assessment

CONTACTS AND LOCATIONS:
Overall Officials: Milena P Mak, MD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo - University of Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mak MP, Pasini FS, Diao L, Garcia FOT, Takahashi TK, Nakazato D, Martins RE, Almeida CM, Kulcsar MAV, Lamounier VA, Nunes EM, de Souza IC, Garcia MRT, Amadio AV, Siqueira SAC, Snitcovsky IML, Sichero L, Wang J, de Castro G Jr. Valproic acid combined with cisplatin-based chemoradiation in locally advanced head and neck squamous cell carcinoma patients and associated biomarkers. Ecancermedicalscience. 2020 Dec 15;14:1155. doi: 10.3332/ecancer.2020.1155. eCollection 2020. PMID 33574900